CLINICAL TRIAL: NCT05536479
Title: Clinical, Radiographic and Histomorphometric Evaluation of Autogenous Stored Versus Autogenous Fresh Mineralized Dentin Graft for Alveolar Ridge Preservation: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Autogenous Stored Versus Autogenous Fresh Mineralized Dentin Graft for Alveolar Ridge Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Wahsh, Principal investigator. Nada Wahsh, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARPerio22
Record Dates: First submitted 2022-09-08; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous stored mineralized dentin graft (ASMDG) (Experimental): Autogenous stored mineralized dentin graft (ASMDG) particles will be prepared by immersing tooth particles in basic ethanol for 10 min for disinfection, then washed twice in saline and dried using sterile gauze The disinfected particles will then be stored at room temperature for 21 days in a sterile container. After 21 days, a second extraction will be performed followed by mixing the stored graft with a few drops of sterile saline to be packed in a socket after extraction
  Interventions: Procedure: Autogenous stored mineralized dentin graft (ASMDG)
- Autogenous fresh mineralized dentin graft (AFMDG) (Active Comparator): Autogenous fresh mineralized dentin graft (AFMDG) particles will be prepared by immersing tooth particles in basic ethanol for 10 min for disinfection, then washed twice in saline and dried using sterile gauze
  Interventions: Procedure: Autogenous fresh mineralized dentin graft (AFMDG)

INTERVENTIONS:
Procedure: Autogenous stored mineralized dentin graft (ASMDG) — Autogenous stored mineralized dentin graft (ASMDG) particles will be prepared by immersing tooth particles in basic ethanol for 10 min for disinfection, then washed twice in saline and dried using sterile gauze.
  The disinfected particles will then be stored at room temperature for 21 days in a sterile container. After 21 days, a second extraction will be performed followed by mixing the stored graft with a few drops of sterile saline to be packed in a socket after extraction
  Arms: Autogenous stored mineralized dentin graft (ASMDG)
Procedure: Autogenous fresh mineralized dentin graft (AFMDG) — Autogenous fresh mineralized dentin graft (AFMDG) particles will be prepared by immersing tooth particles in basic ethanol for 10 min for disinfection, then washed twice in saline and dried using sterile gauze.
  Arms: Autogenous fresh mineralized dentin graft (AFMDG)

SUMMARY:
Tooth extraction triggers a cascade of biological events mediated by both the local inflammatory response that follows the surgical intervention and the deprivation of masticatory stimulation of the periodontium, which elicit an alteration of the homoeostasis and structural integrity of the periodontal tissues. Bone remodeling kicks off after tooth loss and continues for several months with most changes taking place in the first three months.

Interestingly, Schmidt-Schultz and Schultz, found that intact growth factors are conserved even in the collagenous extracellular matrix of ancient human bone and teeth. Thus, the application of stored dentin may have similar benefits as fresh dentin, preserving intact growth factors for a prolonged period avoiding the need to perform multiple surgical interventions simultaneously. The volume of the particulate dentin is more than twice of the original root volume. Thus, the idea of using autogenous stored mineralized dentin grafts (ASMDG) in ARP evolved.

DETAILED DESCRIPTION:
Immediately following tooth extraction, the alveolar ridge comes across its normal physiologic healing process that results in respective alveolar bone loss, structural and compositional changes of the covering soft tissues, as well as morphological alterations.

In an attempt to cutback horizontal and vertical ridge losses, various techniques have been successfully proven to preserve the alveolar ridge including autografts, allografts, xenografts, alloplasts and autogenous dentin grafts. However, fresh autogenous bone graft is still considered gold standard since it exhibits bioactive cell instructive matrix properties and is non-immunogenic and non - pathogenic in spite of the need for harvesting bone and possible morbidity resulting from it. Nevertheless, no gold-standard technique is applicable for every clinical situation.

The similarities between dentin and alveolar bone may help the human body to show an acceptable biological behavior to dentin graft. It is therefore not surprising that dentin that comprises more than 85% of tooth structure can serve as a native bone grafting material, which is reflected by the interaction between mineralized dentin and osteogenic cells that attach and produce mineralized bone matrix directly on the dentin graft.

Mineralized dentin particles have the advantage to maintain its mechanical stability, allowing early loading after grafting in fresh sockets and bone defects where the mineralized dentin is firmly integrated with newly formed bone, creating a solid site for anchorage of dental implants.

Fresh ground dentin has been used successfully as a grafting material alternative in alveolar ridge preservation which has been manifested in that the clinically grafted sites demonstrated limited ridge resorption which allowed for subsequent implant placement without the need to use additional graft biomaterials.

ELIGIBILITY:
Inclusion Criteria:

* Potential candidates requiring extraction of maxillary non-molar teeth.
* Periodontally healthy adjacent teeth.
* Extraction sockets having no more than 50% of buccal alveolar bone loss

Exclusion Criteria:

* Smokers.
* Patients reporting systemic conditions that may compromise healing or bone metabolism (e.g., uncontrolled diabetes, hyperthyroidism).
* Patients having a history of radiotherapy, chemotherapy, or bisphosphonate therapy.
* Females who were pregnant or planning to get pregnant during the study course.
* Root canal treated teeth and teeth with acute infection at the site of extraction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in buccolingual horizontal alveolar ridge width | 4 months
  The horizontal buccolingual alveolar ridge width will be measured radiographically on a CBCT at three levels: at -1 mm, -3 mm, -5 mm below the most coronal aspect of the crest (HW-1, HW-3, HW-5), and clinically by a caliper at -3 mm and -5 mm (HW-3 and HW-5). Measurements will be taken at baseline and after 4 months postoperatively to calculate the change.

SECONDARY OUTCOMES:
Alveolar buccal ridge height | 4 months
  The alveolar buccal ridge height will be measured radiographically on a CBCT at baseline and after 4 months postoperatively.
Postoperative pain | 24 hours
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable')

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Schmidt-Schultz TH, Schultz M. Intact growth factors are conserved in the extracellular matrix of ancient human bone and teeth: a storehouse for the study of human evolution in health and disease. Biol Chem. 2005 Aug;386(8):767-76. doi: 10.1515/BC.2005.090. PMID 16201872